CLINICAL TRIAL: NCT02631941
Title: An Open-Label, Randomized, Five-Period Cross-over, Single-dose Study to Compare Pharmacokinetics Profiles of Z7200 Medium Strength and Symbicort Turbohaler, With and Without Charcoal Blockade in Healthy Volunteers.
Brief Title: Clinical Study to Evaluate Z7200 Pharmacokinetics Profile
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Z7200J04; 2015-003233-95 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Charcoal; Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (10):
- A-B1-B2-C-D (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following 5 treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 days followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B1-C-A-D-B2 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- C-D-B1-B2-A (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- D-B2-C-A-B1 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B2-A-D-B1-C (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- D-C-B2-B1-A (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B2-D-A-C-B1 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- A-B2-B1-D-C (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- B1-A-C-B2-D (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal
- C-B1-D-A-B2 (Experimental): Subjects were dosed on Day 1 of each treatment period with one of the following five treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B2: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal A washout period of a minimum of 5 day followed treatment periods 1 to 4.
  Treatment B1 and B2 denote Symbicort without oral activated charcoal administered in two different period, designated as Symbicort 1 and Symbicort 2.
  Interventions: Drug: Z7200 without oral activated charcoal; Drug: Symbicort Turbohaler without oral activated charcoal; Drug: Z7200 with oral activated charcoal; Drug: Symbicort Turbohaler with oral activated charcoal

INTERVENTIONS:
Drug: Z7200 without oral activated charcoal — 160 ug budesonide and 4.5 ug formoterol fumarate dihydrate, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler (Treatment A).
  Other Names: budesonide/formoterol
Drug: Symbicort Turbohaler without oral activated charcoal — 320 ug budesonide and 9 ug formoterol fumarate dihydrate, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation (Treatments B1 and B2 denote Symbicort without oral activated charcoal administered in two different periods).
  Other Names: budesonide/formoterol
Drug: Z7200 with oral activated charcoal — 160 ug budesonide and 4.5 ug formoterol fumarate dihydrate, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler with a charcoal blockade (Treatment C).
  Other Names: budesonide/formoterol with coadministration of charcoal
Drug: Symbicort Turbohaler with oral activated charcoal — 320 ug budesonide and 9 ug formoterol fumarate dihydrate, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation from a Symbicort Turbohaler, with charcoal blockade (Treatment D).
  Other Names: budesonide/formoterol with coadministration of charcoal

SUMMARY:
Brief Summary:

The primary objective was:

* to assess the bioequivalence of a single dose (two inhalations) of the test product compared to the reference product, with and without charcoal blockade.

The secondary objectives were:

* to assess the pharmacokinetic profile of budesonide and formoterol in plasma after a single dose (two inhalations) of the test product and the reference product, with and without charcoal blockade.
* to assess the safety and tolerability of the test product and the reference product, with and without charcoal blockade.

DETAILED DESCRIPTION:
This was a single center, open label, randomized, five-period crossover, single-dose study in healthy volunteers aged 18 to 45 years. A total of 90 volunteers were planned to be enrolled, with 9 subjects in each of the 10 treatment sequences.

The study consisted of 5 treatment periods, each lasting approximately 48h, separated by a washout period of a minimum of 5 days. RS01 and/or Symbicort Turbohaler device use training was provided on Day -1 and Day 1 of each treatment period. Subjects were screened for eligibility to participate in the study -28 to -2 days prior to the first treatment period, and were randomized to one of 10 treatment sequences containing the following 5 treatment arms on Day 1 of the first treatment period:

Treatment A: Z7200 without oral activated charcoal* Treatment B1: Symbicort 1 without oral activated charcoal* Treatment B2: Symbicort 2 without oral activated charcoal* Treatment C: Z7200 with oral activated charcoal** Treatment D: Symbicort with oral activated charcoal**

Subjects were admitted to the clinical unit at 8.00 on the morning of Day -1, and were dosed on the morning of Day 1 following an overnight fast (minimum of 8h). On Day 2, following collection of the 24-h PK blood sample, subjects were discharged.

* Subjects who received treatments A, B1 and B2 rinsed their mouth vigorously with 50 mL water for 3 to 5 sec immediately after the second inhalation.

** A charcoal blockade was used to prevent absorption from oropharyngeal and GI tract, in order to assess the pulmonary deposition of budesonide and formoterol, with periods performed without a charcoal blockade allowing the assessment of the total systemic exposure to the drug.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female 18 to 45 years of age.
* If female, is currently not pregnant/breast feeding/ or attempting to become pregnant has a negative serum pregnancy test, or is of non-childbearing potential or is of child-bearing potential, willing to commit to using a consistent and acceptable method of birth control or is of child-bearing potential and not sexually active
* Body mass index (BMI) of 18.0 to 32.0 kg/m² inclusive and a body weight ≥50 kg.
* 10 years or more past history of cigarette, <=5 pack year

Main Exclusion Criteria:

* Forced Expiratory Volume in 1 sec (FEV1) value less than 80% of the predicted value and FEV1/FVC (Forced Vital Capacity) ratio <0.7.
* History or current evidence of a clinically significant disease or disorder capable of altering the absorption, metabolism, distribution or elimination of drugs.
* History or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, haematological, neuropsychological, endocrine, gastrointestinal or pulmonary.
* Presence of glaucoma, cataracts, ocular herpes simplex, malignancy, regardless of the clinical significance or current stability of the disease.
* positive tests for Human Immunodeficiency Virus (HIV), Hepatitis B and Hepatitis C.
* Bacterial or viral infection of the upper respiratory tract (including the common cold and flu), sinus, or middle ear within 2 weeks of dosing.
* Lower respiratory tract infection/pneumonia within the past 3 months.
* Presence of any disease or condition or regular concomitant treatment (including vitamins and herbal products) known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Screening haemoglobin value of less than 1g/dL above the Lower Limit of Normality
* History of recurrent vasovagal collapses.
* History of anaphylactic/anaphylactoid reactions.
* History of seizures including febrile seizures excluding childhood febrile convulsions.
* Unable to demonstrate proper inhalation techniques involved in using the delivery devices at screening.
* Exposure to any investigational drug within 90 days of the Screening Visit.
* Known or suspected hypersensitivity or idiosyncratic reaction to any steroid, any β2 agonist; allergy to milk protein.
* Use of an inhaled corticosteroid within 30 days or systemic corticosteroid within 60 days of the Screening Visit.
* Use of medications or herbal medicines that are strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers within 30 days prior to Screening Visit
* Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study.
* Use of caffeine containing beverages more than 5 cups/day.
* Recent or current (suspected) drug abuse or positive result in the drugs abuse test.
* Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 14 units per week for females)
* Predictable poor compliance, intolerance to charcoal solution, or inability to communicate well with the study centre personnel or inability to participate in all treatment periods.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, Principal Investigator — Quotient Clinical Limited
Locations (1):
- Quotient Clinical Ltd, Ruddington, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened for eligibility -28 to -2 days prior to the first treatment period. On Day -1 of the first treatment period, i.d. before randomization, subjects were trained on both the RS01 and Symbicort Turbohaler devices.
Pre-assignment Details: Subjects had to have an adequate inspiratory flow rate and be able to use both inhalers. Subjects who continued to meet all entry criteria on Day -1 of treatment Period 1 and with an inspiratory flow rate of ≥60 L/min and proper device use entered the treatment phase.
Groups:
- A-B1-B2-C-D; B1-C-A-D-B2; C-D-B1-B2-A; D-B2-C-A-B1; B2-A-D-B1-C; D-C-B2-B1-A; B2-D-A-C-B1; A-B2-B1-D-C; B1-A-C-B2-D; C-B1-D-A-B2: Subjects were dosed on Day 1 of each treatment period with one of the following 5 treatments according to the randomization schedule using a Williams Latin Square design:
  1. Treatment A: Z7200 without oral activated charcoal
  2. Treatment B1: Symbicort 1 without oral activated charcoal
  3. Treatment B1: Symbicort 2 without oral activated charcoal
  4. Treatment C: Z7200 with oral activated charcoal
  5. Treatment D: Symbicort with oral activated charcoal
  A washout period ≥5 days followed treatment periods 1 to 4.
  Z7200 without activated charcoal: 160 ug budesonide and 4.5 ug formoterol, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler (Treatment A).
  Symbicort Turbohaler without activated charcoal: 320 ug budesonide and 9 ug formoterol, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation (Treatments B1 and B2).
  Z7200 with activated charcoal: 160 ug budesonide and 4.5 ug formoterol, administered as two inhalations (2 x Z7200 capsules) of budesonide 80 ug/inhalation and formoterol 2.25 ug/inhalation, using an RS01 inhaler with a charcoal blockade (Treatment C).
  Symbicort Turbohaler with activated charcoal: 320 ug budesonide and 9 ug formoterol, administered as two inhalations of budesonide 160 ug/inhalation and formoterol 4.5 ug/inhalation, with charcoal blockade (Treatment D).
Period: Overall Study
Arm/Group | A-B1-B2-C-D | B1-C-A-D-B2 | C-D-B1-B2-A | D-B2-C-A-B1 | B2-A-D-B1-C | D-C-B2-B1-A | B2-D-A-C-B1 | A-B2-B1-D-C | B1-A-C-B2-D | C-B1-D-A-B2
Started | 9 | 10 | 9 | 9 | 9 | 8 | 9 | 9 | 10 | 9
A | 9 | 8 | 9 | 9 | 9 | 8 | 9 | 9 | 9 | 9
B1 | 9 | 10 | 9 | 9 | 8 | 8 | 9 | 9 | 10 | 9
B2 | 9 | 8 | 9 | 9 | 9 | 8 | 9 | 9 | 9 | 9
C | 9 | 8 | 9 | 9 | 8 | 8 | 9 | 8 | 9 | 9
D | 9 | 8 | 9 | 9 | 8 | 8 | 9 | 9 | 9 | 9
Completed | 9 | 8 | 9 | 9 | 8 | 8 | 9 | 8 | 9 | 9
Not Completed | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All subjects who received at least one dose (2 inhalations) of investigational medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | A-B1-B2-C-D | B1-C-A-D-B2 | C-D-B1-B2-A | D-B2-C-A-B1 | B2-A-D-B1-C | D-C-B2-B1-A | B2-D-A-C-B1 | A-B2-B1-D-C | B1-A-C-B2-D | C-B1-D-A-B2 | Total
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 9 | 8 | 9 | 9 | 10 | 9 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 9 | 9 | 9 | 8 | 9 | 9 | 10 | 9 | 91
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (8.1) | 29.9 (9.0) | 32.9 (9.4) | 30.8 (8.3) | 23.8 (3.8) | 26.1 (8.5) | 25.8 (6.9) | 31.7 (7.7) | 30.7 (9.7) | 26.2 (7.2) | 28.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 2 | 4 | 2 | 1 | 3 | 3 | 1 | 29
  Male | 5 | 5 | 5 | 7 | 5 | 6 | 8 | 6 | 7 | 8 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 4
  White | 6 | 9 | 9 | 8 | 6 | 7 | 8 | 8 | 7 | 9 | 77
  More than one race | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 10 | 9 | 9 | 9 | 8 | 9 | 9 | 10 | 9 | 91

OUTCOME MEASURES:

1. Primary Outcome: AUC0-last of Budesonide With and Without Charcoal Blockade
Description: Area under the plasma concentration-time curve from time zero to the last detectable level calculations were performed using the linear trapezoidal rule. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: PK population included subjects who had received both test and reference for at least one dose of each treatment without or with oral charcoal.
  Treatment B "Number of Participants" counted for both Symbicort 1 and Symbicort 2 treatment group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Treatment A: Z7200 without charcoal (160 ug budesonide)
- Treatment B: Symbicort 1+2 without charcoal (320 ug budesonide)
- Treatment C: Z7200 with charcoal (160 ug budesonide)
- Treatment D: Symbicort with charcoal (320 ug budesonide)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
pg*h/mL | 1710 (17.9) | 1710 (33.1) | 1570 (20.2) | 1530 (39.7)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — For budesonide AUC0-last, the 90% Cls for Z7200 compared with Symbicort without and with charcoal lie entirely within the standard bioequivalence acceptance limits of (80% - 125.00%); p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 100.64, 90% CI 2-sided [95.82 to 105.69]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Adjusted geometric means ratio = 102.11, 90% CI 2-sided [95.55 to 109.13]

2. Primary Outcome: AUC0-last of Formoterol With and Without Charcoal Blockade
Description: as for outcome 1
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
pg*h/mL | 46.1 (22.7) | 52.6 (37.3) | 39.0 (25.4) | 42.8 (50.8)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — For Formoterol AUC0-last, the 90% Cls for Z7200 compared to Symbicort without and with charcoal lie entirely within the standard bioequivalence acceptance limits of (80.00%, 125.00%); p = 0.002, Mixed Models Analysis; Adjusted geometric means ratio = 87.96, 90% CI 2-sided [83.31 to 92.86]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.005, Mixed Models Analysis; Adjusted geometric means ratio = 91.17, 90% CI 2-sided [83.94 to 99.04]

3. Primary Outcome: Cmax of Budesonide With and Without Charcoal Blockade
Description: Maximum plasma level of budesonide with and without charcoal blockade. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
pg/mL | 1080 (69.8) | 686 (53.2) | 1110 (72.8) | 663 (50.6)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — For Budesonide Cmax, the 90% Cls for Z7200 compared with Symbicort without and with charcoal do not lie entirely within the wider bioequivalence acceptance limits of ( 73.74%, 135.62%) and standard bioequivalence acceptance limits of (80.00%, 125.00%), respectively; p = 1.00, Mixed Models Analysis; Adjusted geometric means ratio = 157.86, 90% CI 2-sided [144.12 to 172.91]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 1.00, Mixed Models Analysis; Adjusted geometric means ratio = 166.81, 90% CI 2-sided [148.35 to 187.57]

4. Primary Outcome: Cmax of Formoterol With and Without Charcoal Blockade
Description: Maximum plasma level of formoterol with and without charcoal blockade. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
pg/mL | 10.1 (37.1) | 11.9 (46.1) | 10.3 (35.7) | 11.7 (50.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — For Formoterol Cmax, the 90% Cl for Z7200 compared to Symbicort without and with charcoal lie entirely within the wider bioequivalence acceptance limits of (77.65%, 128.79%) and standard bioequivalence acceptance limits of (80.00%, 125.00%), respectively; p = 0.012, Mixed Models Analysis; Adjusted geometric means ratio = 85.22, 90% CI 2-sided [79.66 to 91.17]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.020, Mixed Models Analysis; Adjusted geometric means ratio = 87.74, 90% CI 2-sided [81.48 to 94.47]

5. Secondary Outcome: AUC0-30 of Budesonide With and Without Charcoal Blockade.
Description: Area under the plasma concentration-time curve from time zero to 30 minutes calculations were performed using the linear trapezoidal rule. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-30 min (0, 2, 5, 10, 15, 20, and 30 min)
Population: PK population included subjects who had received both test and reference for at least one dose of each treatment without or with oral charcoal.
  Treatment B "Number of Participants" counted for both Symbicort 1 and Symbicort 2 treatment groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
pg*h/mL | 313 (30.5) | 238 (48.9) | 315 (32.5) | 237 (47.5)

6. Secondary Outcome: AUC0-30 of Formoterol With and Without Charcoal Blockade.
Description: as for outcome 5
Time Frame: 0-30 min (0, 2, 5, 10, 15, 20, and 30 min)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
pg*h/mL | 3.37 (30.1) | 3.88 (42.1) | 3.36 (29.7) | 3.76 (47.9)

7. Secondary Outcome: AUC0-∞ of Budesonide With and Without Charcoal Blockade
Description: Area under the plasma concentration-time curve from time zero to infinity calculations were performed using the linear trapezoidal rule. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 171 | 85 | 85
pg*h/mL | 1820 (18.2) | 1830 (33.0) | 1670 (20.3) | 1640 (38.5)

8. Secondary Outcome: AUC0-∞ of Formoterol With and Without Charcoal Blockade
Description: as for outcome 7
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 163 | 84 | 79
pg*h/mL | 55.4 (23.4) | 63.0 (36.0) | 46.8 (26.1) | 53.7 (37.6)

9. Secondary Outcome: Tmax for Budesonide With and Without Charcoal Blockade
Description: Time at which the maximum plasma level (Cmax) occurred with and without charcoal blockade. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
hours | 0.080 [0.03 to 0.51] | 0.250 [0.03 to 1.00] | 0.040 [0.03 to 0.75] | 0.250 [0.03 to 1.00]

10. Secondary Outcome: Tmax for Formoterol With and Without Charcoal Blockade
Description: as for outcome 9
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 172 | 86 | 86
hours | 0.080 [0.04 to 0.25] | 0.080 [0.03 to 0.33] | 0.080 [0.08 to 0.25] | 0.080 [0.08 to 0.51]

11. Secondary Outcome: t1/2 for Budesonide With and Without Charcoal Blockade
Description: Apparent elimination half-life calculated as 0.693/lambda zeta, with and without charcoal blockade. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 87 | 171 | 85 | 85
hours | 3.21 (22.2) | 3.14 (23.2) | 3.23 (23.6) | 3.01 (23.4)

12. Secondary Outcome: t1/2 for Formoterol With and Without Charcoal Blockade
Description: as for outcome 11
Time Frame: 0-24h (0, 2, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 1440 min)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 83 | 163 | 84 | 79
hours | 9.35 (25.4) | 9.28 (26.6) | 9.45 (27.6) | 9.08 (26.8)

13. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 refers to the volume of air that an individual can exhale during a forced breath in 1 second. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: At 75 min (1.25 hours) post-dose
Population: Safety population: all subjects who received at least one dose (2 inhalations) of investigational medicinal product Treatment B "Number of Participants" counted for both Symbicort 1 and Symbicort 2 treatment groups.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 88 | 91 | 86 | 87
liters | 0.188 (0.167) | 0.170 (0.161) | 0.173 (0.143) | 0.153 (0.131)

14. Secondary Outcome: Change From Baseline in the Ratio of Forced Expiratory Volume in 1 Second to Forced Vital Capacity (FEV1/FVC)
Description: FVC = Forced vital capacity. It is the full amount of air that can be exhaled with effort in a complete breath.
  FEV1/FVC = Tiffenau-Pinelli Index. This parameter represents the measurement of the amount of air an individual can forcefully exhale from his/her lungs. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: At 75 min (1.25 hours) post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 88 | 91 | 86 | 87
Ratio | 3.94 (3.72) | 3.78 (2.90) | 3.75 (2.73) | 3.83 (2.84)

15. Secondary Outcome: Change From Baseline in Peak Expiratory Flow Rate (PEFR)
Description: PEFR is the highest rate at which gases can be expelled from the lungs via an open mouth. Its measurement is a simple procedure in which an individual takes a full inspiration and blows out as forcibly as possible into an instrument called a peak flow meter, which measures the maximal gas flow in an exhalation in liters per minute. Participants for the Treatment B are counted for both Symbicort 1 and Symbicort 2, together.
Time Frame: At 75 min (1.25 hours) post-dose
Population: Safety population: all subjects who received at least one dose (2 inhalations) of investigational medicinal product.
  Treatment B "Number of Participants" counted for both Symbicort 1 and Symbicort 2 treatment groups.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 88 | 91 | 86 | 87
L/min | 32.3 (42.0) | 22.4 (38.7) | 30.3 (34.3) | 19.3 (39.1)

ADVERSE EVENTS:
Time Frame: Throughout the study till the end of trial assessment, that is from the first day of screening up to 6 weeks.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/91 | 0/86 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/91 | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 15/88 | 22/91 | 13/86 | 11/87
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=88) | Treatment B (N=91) | Treatment C (N=86) | Treatment D (N=87)
Headache (Nervous system disorders) | 5 (6) | 6 (7) | 6 (6) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (4) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site rash (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoasthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations and Caveats not specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No